CLINICAL TRIAL: NCT01269775
Title: Comparison of Face to Face Lecture Based, Interactive Internet Based and Computer Based Teaching Regarding Students' Knowledge Achievement and Satisfaction: A Randomized Controlled Trial
Brief Title: Comparison of Face to Face Lecture, Interactive Internet Based and Computer Based Teaching
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Aeen Mohammadi, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 10764
Record Dates: First submitted 2011-01-02; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: 3rd Year Medical School's Students

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Face to face lecture (Experimental): The lecturer allocated 1.5 hours for delivering the lecture by using provided slides about the topic and 0.5 hours for question and answer.
  Interventions: Other: Teaching Methods
- Internet based teaching (Experimental): For providing materials for interactive internet-based group the professor's lecture was converted to an interactive electronic content. This content started with a case introduction followed with asking questions and then based on each student's answer a learning pathway would be assigned to his/her.
  Interventions: Other: Teaching Methods
- Computer based teaching (Experimental): For providing material for computer-based group the lecture of the same professor was recorded in studio environment and was synchronized with the slides that were similar to those for lecture-based group. Then the lecture and the slides were converted to a CD as a multimedia CD.
  Interventions: Other: Teaching Methods

INTERVENTIONS:
Other: Teaching Methods — We carried out a randomized controlled trial comparing three methods of teaching. These three instructional methods consist of face to face lecture, interactive internet based teaching and computer based teaching (lecture synchronized with presentation) regarding medical students' knowledge achievement and satisfaction.

SUMMARY:
The investigators carried out a randomized controlled trial comparing three methods of teaching. These three instructional methods consist of face to face lecture, interactive internet based teaching and computer based teaching (lecture synchronized with presentation).

The hypotheses tested were: a) whether there is a difference between these three methods in knowledge achievement and b) whether there is a difference between Students satisfaction in three groups.

ELIGIBILITY:
Inclusion Criteria:

* 3rd year medical school's students

Exclusion Criteria:

* It must be their first experience of the course and they must have no previous elective or obligatory study about teaching topic (multiple myeloma).

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 84
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aeen Mohammadi, Instructor, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran